CLINICAL TRIAL: NCT01360710
Title: The Effect of Moxonidine and Regression of Early Target Organ Damage in Young Subjects With Abdominal Obesity and Hypertension: a Randomised, Double Blind, Active Comparator Clinical Trial
Brief Title: The Effect of Moxonidine on Blood Pressure and Regression of Early Target Organ Damage in Young Subjects With Abdominal Obesity and Hypertension
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baker Heart and Diabetes Institute (Other)
Responsible Party: Principal Investigator, Markus Schlaich, A/Prof, Baker Heart and Diabetes Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Young obese hypertension
Record Dates: First submitted 2011-05-24; First posted 2011-05-26 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Abdominal Obesity; Hypertension
Keywords: male age 18-30 years old; presence of central obesity; no history of cardiovascular disease, depression; not on any medication
MeSH Terms: conditions — Obesity, Abdominal; Hypertension; Depression | interventions — moxonidine; Irbesartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Moxonidine (Experimental)
  Interventions: Drug: Moxonidine
- Irbesartan (Active Comparator)
  Interventions: Drug: Irbesartan

INTERVENTIONS:
Drug: Moxonidine — 0.2mg/day for 2 weeks, 0.4mg/day for 6 months
  Other Names: Brand name = Physiotens
  Arms: Moxonidine
Drug: Irbesartan — 75 mg/day for 2 weeks and then 150 mg/day for 24 weeks.
  Arms: Irbesartan

SUMMARY:
Obesity is a major risk factor for the development of hypertension. Based on population studies, risk estimates indicate that at least two-thirds of the prevalence of hypertension can be directly attributed to obesity. Obesity per se is commonly associated with activation of the sympathetic nervous system with a predominant increase in sympathetic outflow to the kidneys and the peripheral vasculature and there is now conclusive evidence that heightened sympathetic nerve activity is a major contributor to the elevation in blood pressure associated with obesity, particularly in young subjects. In line with these findings, dietary weight loss has repeatedly been demonstrated to result in reduced sympathetic nerve activity and lower blood pressure levels.

Several lines of evidence have well documented the significant role of SNS activation in obesity associated hypertension and target organ damage. Weight loss is the preferred treatment option for obesity and its consequences and reduces both SNS activation and blood pressure. In the real world however, weight loss maintenance is rarely achieved in obese patients highlighting the urgent need for alternative treatment strategies. Given the crucial involvement of SNS activation in various aspects of the obesity related increase in blood pressure, target organ damage and cardiovascular risk, the use of sympatho-inhibitory agents at an early stage is an obvious choice.

The investigators therefore plan to examine the effects of the centrally sympatholytic agent moxonidine on blood pressure and the morning surge in blood pressure, sympathetic activity, regression of early target organ damage (heart, kidney and endothelium), metabolic and inflammatory markers in young obese subjects with hypertension in a randomized, double-blind clinical trial with the angiotensin receptor blocker irbesartan as an active comparator to achieve similar blood pressure reductions in both groups. The investigators hypothesize that moxonidine treatment will result in significant improvements in these outcome parameters and beneficial effects beyond simple blood pressure reduction.

Findings from this study could pave the way for an early and pathophysiology- tailored treatment strategy of obesity related hypertension and its detrimental consequences.

ELIGIBILITY:
Inclusion Criteria:

* male age 18-30 years old
* presence of central obesity and hypertension
* no history of cardiovascular disease or depression
* not on any medication

Exclusion Criteria:

* history of cardiovascular disease, depression or anxiety disorder

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Microneurography (nerve recording) | 6 months
  Microneurography technique will be performed on participants at baseline and 6 months post treatment to see if moxonidine has any effect in the reduction of sympathetic activiry.

SECONDARY OUTCOMES:
Blood test | 6 months
  Blood samples will be taken from antecubital vein for biochemical analyses purposes. The sampling will take place at baseline and at 6 months visit.

CONTACTS AND LOCATIONS:
Locations (1):
- BakerIDI Heart and Diabetes Institute, Prahran, Victoria, Australia